CLINICAL TRIAL: NCT01219946
Title: A Cross Sectional Study for the Assessment of the Words Used by Patients and Physicians to Express the Symptoms of Chronic Obstructive Pulmonary Disease and the Limitations of Patients' Activities in Primary Care.
Brief Title: A Study for the Assessment of the Words Used by Patients and Physicians to Express the Symptoms of Chronic Obstructive Pulmonary Disease (COPD)
Acronym: COPD Language
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RGR-DUM-2010/1
Record Dates: First submitted 2010-10-08; First posted 2010-10-13 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease, symptoms
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Chronic Obstructive Pulmonary Disease

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is characterized by a progressive decline in lung function and increased symptoms such as breathlessness/dyspnoea, cough and expectoration.

Even though subjective in nature, the symptomatology of COPD and mainly that of breathlessness/dyspnoea has been studied with the use of objective measurement tools. Taking into consideration that the symptoms experienced by the patient who suffers from a progressive disease such as COPD can only be perceived and interpreted by the patient him- or herself, and thus difficult to be quantified, COPD remains a challenge in clinical research.

Therefore, there is a need to carry out qualitative studies that will provide insight into the wide spectrum of COPD symptomatology from the patient's perspective. In addition, a further mapping of the impact that COPD symptoms' perception has on a patient's life is required, as well as of the different pathways through which symptoms' perception is interpreted regarding the limitations of daily living activities, and the subsequent impact on disease management. The more the physician learns on the embodied experience of COPD, the better he/she may assist the patient in achieving optimal COPD management.

Thus this cross-sectional observational study was designed aiming to obtain these data. Specifically, the study aims to evaluate the most frequently used words by the patients and the physicians to express the symptoms of COPD as well as the limitation of activities that it causes.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-75 years
* Current or former smokers
* Known history of COPD for at least 6 months before enrolment into the study documented by spirometry (FEV1 /FVC <70%)
* Patients with stable COPD (no exacerbation within the last month before enrolment into the study) under treatment with a long-acting inhaled bronchodilator (LABA and/or LAMA) alone or in combination with an inhaled corticosteroid
* Written consent for participation in the study
* Patients who are able to complete by themselves in Greek a questionnaire on COPD.

Exclusion Criteria:

* Patients with diagnosed Asthma
* Patients with any psychiatric, neurological or other disorder render them unable to complete the COPD questionnaire by themselves
* The patient participates in another study.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Obstructive Pulmonary Disease
Sampling Method: Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Words used by the patients and the physicians to express the symptoms of COPD as well as the limitations of patients' daily living activities caused by COPD. | End of recruitment (estimated timeframe :2.5 months)

SECONDARY OUTCOMES:
Age | End of recruitment (estimated timeframe :2.5 months)
Gender | End of recruitment (estimated timeframe :2.5 months)
Place of residence | End of recruitment (estimated timeframe :2.5 months)
Marital status | End of recruitment (estimated timeframe :2.5 months)
Native language | End of recruitment (estimated timeframe :2.5 months)
Educational level | End of recruitment (estimated timeframe :2.5 months)
Occupation | End of recruitment (estimated timeframe :2.5 months)
Co-morbidities | End of recruitment (estimated timeframe :2.5 months)
Years / months since COPD diagnosis and years with COPD symptoms | End of recruitment (estimated timeframe :2.5 months)
Smoking history | End of recruitment (estimated timeframe :2.5 months)
Number of exacerbations during the last year | End of recruitment (estimated timeframe :2.5 months)
Current therapy | End of recruitment (estimated timeframe :2.5 months)
CCQ score | End of recruitment (estimated timeframe :2.5 months)
Compliance with therapy | End of recruitment (estimated timeframe :2.5 months)
Actions/therapeutic recommendations by the physician associated with each chosen word that express the chronic daily symptoms | End of recruitment (estimated timeframe :2.5 months)
Scale for the assessment of the severity of the relevant symptoms | End of recruitment (estimated timeframe :2.5 months)
Actions/therapeutic recommendations by the physician when any of the symptoms worsen | End of recruitment (estimated timeframe :2.5 months)
Severity scale regarding how the patient experiences each of the chosen words that express the chronic daily symptoms | End of recruitment (estimated timeframe :2.5 months)
Related actions initiated by the patient regarding chronic daily symptoms | End of recruitment (estimated timeframe :2.5 months)
Related actions initiated by the patient when the symptoms worsen. | End of recruitment (estimated timeframe :2.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, Study Director
Locations (32):
- Greece (32):
  - Research Site, Athens, Attica
  - Research Site, Kallithea, Attica
  - Research Site, Marousi, Attica
  - Research Site, Megara, Attica
  - Research Site, Nea Ionia, Attica
  - Research Site, Nea Makri, Attica
  - Research Site, Piraeus, Attica
  - Research Site, Chania, Crete
  - Research Site, Heraklion, Crete
  - Research Site, Rhodes, Dodekanisa
  - Research Site, Corfu, Eptanisa
  - Research Site, Ioannina, Ipiros
  - Research Site, Larissa, Kyklades
  - Research Site, Mykonos, Kyklades
  - Research Site, Alexándreia, Makedonia
  - Research Site, Drama, Makedonia
  - Research Site, Florina, Makedonia
  - Research Site, Katerini, Makedonia
  - Research Site, Kavala, Makedonia
  - Research Site, Kozani, Makedonia
  - Research Site, Serres, Makedonia
  - Research Site, Thesaloniki, Makedonia
  - Research Site, Krestena, Peloponisos
  - Research Site, Lechainá, Peloponisos
  - Research Site, Pátrai, Peloponisos
  - Research Site, Skála, Peloponisos
  - Research Site, Agrinio, Sterea
  - Research Site, Halkida, Sterea
  - Research Site, Itea, Sterea
  - Research Site, Livadia, Sterea
  - Research Site, Volos, Thesalia
  - Research Site, Xánthi, Traki